CLINICAL TRIAL: NCT06755606
Title: Evaluation of the Effect of an Emergency Department Information Video on the Risk of Post-Traumatic Stress Disorder 30 Days After an Emergency Visit.
Acronym: VISU
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231231; IDRCB : 2023-A01766-39 (Other: ANSM)
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: PTSD - Post Traumatic Stress Disorder; Stress Disorder, Post Traumatic
Keywords: stress disorders; interventions; communication; emergency medicine
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- BEFORE: Group pf patients enrolled Before the information procedure was set up
- AFTER: Group pf patients enrolled After the information procedure was set up

SUMMARY:
Post-traumatic stress disorder (PTSD) is a psychological disorder characterized by the re-experiencing of distressing symptoms, avoidance of traumatic memories and physiological hyperarousal in people who have been exposed to a traumatic event. The consequences of PTSD are manifold: financial, quality of life, absenteeism, morbidity, and mortality.

An emergency department visit can be a traumatic event and associated with anxiety.

Studies have explored the prevalence and factors associated with the occurrence of PTSD among a selected population of patients admitted to the emergency department for either cardiological or traumatological reasons. The prevalence of PTSD at 1 month varied among these populations, from 12% to 25%.

Several factors have been described that could be independently associated with an increased risk of developing PTSD: factors linked to the patient himself (basal state and severity of acute pathology) or to the patient pathway (care structure, care modalities, waiting time). Given the serious medical, psycho-social and economic consequences of PTSD, it is important to identify the risk factors that can be controlled during a patient's stay in the emergency department.

In 2025, a general information procedure for patients and next of kin will be deployed in three emergency departments.

The aim of this procedure is to improve the quality of the information provided to emergency patients, thereby enhancing the experience of patients and those accompanying them. It will consist of video support delivering standardized information to patients from the moment they arrive in the emergency department until they are discharged. These videos will describe the patient's journey through the emergency department.

The aim of this study is to evaluate the effect of this information procedure on the risk of developing PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Triage level 1, 2, 3 by the triage nurse (according to CIMU, FRENCH or other scale used locally)
* Non-opposition to participation in the study after information and delivery of the information note
* Possibility of 30-day follow-up (self-questionnaire to be completed by e-mail)
* Patient with cognitive or sensory capacity to view and understand information videos

Exclusion Criteria :

* Inability to consent (neurological disorder, coma, acute intoxication, cognitive impairment)
* Patient does not have a good understanding of the French language.
* Estimated life expectancy less than 6 months
* Participation in other clinical intervention research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient coming for an unscheduled emergency consultation
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Occurence PTSD | DaAy 30
  assessed by calculation of PCL-5 score

SECONDARY OUTCOMES:
Identify factors associated with the occurrence of PTSD | Day 30
  Identify factors associated with the occurrence of PTSD in relation to the acute pathology, the patient's baseline condition, and the patient's pathway through the emergency department.
HAD score at D30 | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer TRUCHOT, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Undecided